CLINICAL TRIAL: NCT05421507
Title: A Serial Case, Single-arm, Real-world Study of the Safety and Efficacy of 3D-printed Coplanar Template Combined With CT-guided Radioactive I-125 Seed Implantation in the Treatment of Head and Neck Tumors
Brief Title: 3D-PCT Combined With CT-guided Radioactive I-125 Seed Implantation in the Treatment of Head and Neck Tumors
Status: Recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Qiu Bin, Principe Investigator, Peking University Third Hospital
Other Study IDs: CHiECRCT20220018
Record Dates: First submitted 2022-05-24; First posted 2022-06-16 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Malignant Tumor of Head and/or Neck
Keywords: iodine-125 seeds implantation; 3D printing non co-planar template; Malignant Tumor of Head and/or Neck
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with head and neck tumors with local recurrence or metastasis: The patients in the group were treated with routine clinical treatment: 3D-PCT combined with CT-guided I-125 seeds implantation in the treatment of head and neck malignant tumors.
  The prescription dose is given 110-150Gy according to tumor pathological type, tumor volume, history of previous radiotherapy and different surrounding normal tissues according to experience and routine diagnosis and treatment.
  Interventions: Radiation: Radioactive Iodine-125 Seeds Implantation

INTERVENTIONS:
Radiation: Radioactive Iodine-125 Seeds Implantation — Radioactive Iodine-125 Seeds Implantation(RISI) belongs to permanent inter-tissue brachytherapy. Guided by CT or ultrasound,radioactive I-125 seeds are implanted into tumor tissue, and radioactive I-125 continuously releases radiation to kill tumor cells.Radioactive I-125 seeds can reach a higher dose in the tumor, and the dose of the normal tissue around the tumor is lower, and the damage to the normal tissue is less while reaching the radical dose. The NCCN guidelines recommend RISI as the standard treatment for early prostate cancer. For early prostate cancer, RISI can achieve comparable efficacy as surgery, complications and side effects are lower than surgery, therefore patients can obtain better quality of life. RISI is also recommended by NCCN as one of the treatments for locally recurrent rectal cancer. Several studies have confirmed that RISI is safe and effective in the treatment of locally advanced or recurrent head and neck, chest, abdominal and retroperitoneal tumors.

SUMMARY:
The purpose of this study is to verify the accuracy, short-term efficacy and side effects of 3D printing coplanar template combined with CT-guided I-125 seeds implantation in the treatment of malignant tumors of the head and neck.

DETAILED DESCRIPTION:
Iodine-125 seeds Implantation (RISI) for the treatment of tumors, mainly with the help of imaging guidance, the radioactive I-125 seeds radioactive source is directly implanted into the tumor tissue, and the purpose of killing tumor cells is achieved through the continuous release of radiation by radionuclide. At present, it has been clinically used in the local treatment of tumors in head and neck, chest, abdomen, pelvis, spine, columns and limbs. The main technical difficulties in implementing RISI lies in the complexity of operation and the control of operation quality.In the era of unarmed puncture, the quality of operation is difficult to guarantee, and the therapeutic effect is quite different.In 2015, our unit carried out RISI technology under the guidance of 3D model plates, which significantly improved the treatment accuracy of RISI.

The current 3D printing templates are divided into two types: non-coplanar template (3D-PNCT) and coplanar template (3D-PCT). In clinical practice, due to the complex technical requirements, high production cost and long printing time of non-coplanar mold board, a considerable number of patients can be well treated with coplanar template.Compared with the non-coplanar individualized template, the coplanar template has the advantages of accurate needle path control, rapid needle path adjustment, convenient real-time optimization, batch production without waiting for template printing time, and the operation is easy to process, easy for doctors to grasp quickly, the cost is lower than non-coplanar template, and easy to carry out at the grass-roots level. However, most of the existing clinical application data of the template come from the non-coplanar template, and the dosimetry, needle path error and clinical effect of particle implantation guided by the coplanar template are still lack of research. Therefore, this study intends to explore the coplanar template technology and analyze the safety and effectiveness of 3D printing coplanar template combined with CT-guided I-125 seeds implantation in the treatment of head and neck malignant tumors.

The purpose of this study is to verify the accuracy, short-term efficacy and side effects of 3D printing coplanar template combined with CT-guided I-125 seeds implantation in the treatment of malignant tumors of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

* the age is 18-80 years old;
* the pathological diagnosis is clear, patients with local recurrence / metastasis of head and neck tumor after operation or external radiotherapy;
* the tumor diameter ≤ 5cm, the number of lesions ≤ 3;
* there is a suitable puncture path, and the target dose of pre can reach the prescribed dose;
* KPS ≥ 70 points, the expected survival time is more than 3 months;
* patients have signed a consent form for I-125 seeds implantation therapy;
* patients have signed the consent form of knowing emotions to participate in this observational study;

Exclusion Criteria:

* coagulation dysfunction;
* tumor surface rupture, or tumor memory liquefied and necrotic in a large range, with poor expected particle distribution;
* severe underlying diseases, resulting in unsafe completion of I-125 seeds implantation therapy, including active infections requiring drug treatment;
* mental abnormalities affecting cognitive ability;
* poor compliance and inability to complete treatment;
* those who were considered unsuitable to participate in this clinical trial;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size was calculated by One-Sample Log-rank Tests in PASS 15 software. Class I error probability (α) = 0. 05; class II error probability (β) = 0. 2, that is, power = 1-β = 0. 8. According to the experience and data of the center, it is assumed that the local control index can be more than doubled by reducing RISI, that is, Hazard Rates113 (M1:M0) = 2:1. Finally the sample size was calculated to be 25 cases, and the sample size of was estimated to be 30 cases considering the 20% loss of follow-up rate.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-05-28 (Estimated); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Adverse events(operation-related complications and radiation side effects) | The side effects were completely observed after 2 years of follow-up.The follow-up interval was calculated from the completion of the treatment, once every 3 months in the first year and once every 6 months in the second year.
  Adverse events are commonly used in the term v5.0 to evaluate the side effects after treatment. The evaluation organ depends on the specific condition of the treatment site and the tissue adjacent to the target area. Other adverse events included particle displacement, needle implantation transfer, and operation-related complications (bleeding, nerve injury, etc).

SECONDARY OUTCOMES:
Local progression free survival | The local progression free survival were completely observed after 2 years of follow-up.The follow-up interval was calculated from the completion of the treatment, once every 3 months in the first year and once every 6 months in the second year.
  The length of time during and after the treatment of the head and neck tumors, that a patient lives with the disease but it does not get worse.
Overall survival | he overall survival were completely observed after 2 years of follow-up.The follow-up interval was calculated from the completion of the treatment, once every 3 months in the first year and once every 6 months in the second year.
  Overall survival (OS) is defined as the time from follow up to death.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiation Oncology of Peking university third hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No